CLINICAL TRIAL: NCT00635544
Title: Healthy Life Style in Europe by Nutrition in Adolescence: Cross-Over Multicentre Study
Brief Title: Cross-Over Multicentre Study in Adolescents
Acronym: HELENA-COMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Prof Luca Scalfi, University of Napoli "Federico II"
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: H3; Contract number: 007034
Record Dates: First submitted 2008-03-06; First posted 2008-03-13 (Estimated); Last update posted 2009-01-28 (Estimated); Status verified 2009-01

CONDITIONS: Overweight; Hyperlipidemia
Keywords: Adolescence; Overweight; Dietary Fiber; Glycemic Index; Healthy lifestyle
MeSH Terms: conditions — Overweight; Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): dietary treatment with a high-glycemic index low-fibre diet (HGI-LF)
  Interventions: Other: dietary treatment
- 2 (Active Comparator): dietary treatment with a low-glycemic index high-fibre diet (LGI-HF)
  Interventions: Other: dietary treatment

INTERVENTIONS:
Other: dietary treatment — dietary treatment with a high-glycemic index low-fibre diet (HGI-LF)
  Arms: 1
Other: dietary treatment — dietary treatment with a low-glycemic index high-fibre diet (LGI-HF)
  Arms: 2

SUMMARY:
The main objective of this study is to evaluate the effects of two diets with different glycemic index and fibre content on glucose metabolism and plasma lipid profile of 80 adolescents in 4 European centres.

Secondary objectives are to evaluate the effects of the two standardized diets on selected hormones and variables linked to inflammatory status.

ELIGIBILITY:
Inclusion Criteria:

* Age 13-16 yrs
* Written informed consent
* Menstrual cycle for at least 6 months
* Overweight

Exclusion Criteria:

* Taking part simultaneously in another research trial
* Involvement in physical training (>4 h/week of vigorous physical activity)
* Any dietary treatment in the previous two months
* Body weight changes > 3 kg in the previous two months
* Gastrointestinal diseases, irritable bowel syndrome, or positive history for recurrent gastrointestinal symptoms such as nausea, vomiting, bloating, epigastric pain, abdominal pain, abdominal discomfort, flatulence, severe constipation
* Kidney diseases
* Type 1 or type 2 diabetes
* Thyroid or other hormonal diseases
* Other secondary causes (including illnesses) of hyperlipidemia or altered glucose metabolism
* Severe hyperlipidemia (total cholesterol > 300 mg/dL or triglycerides >300 mg/dL)
* Severe hypertension
* Positive history for eating disorders
* Any regular drug treatment
* Any food allergy and intolerance

Ages: 13 Years to 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2007-01; Primary Completion 2008-01 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
blood glucose and lipids | after 3 weeks of dietary treatment

SECONDARY OUTCOMES:
blood hormones and inflammatory status parameters | after 3 weeks of dietary treatment

CONTACTS AND LOCATIONS:
Locations (4):
- Department of Nutrition and Dietetics, Harokopio University, Athens, Greece
- Pécsi Tudományegyetem Anyagcseregondozó, Pécs, Hungary
- Dipartimento di Pediatria Università di Napoli "Federico II", Napoli, Italy
- Instituto del Frio. Departamento de Metabolismo y Nutrición, Madrid, Spain

REFERENCES:
- See also: HELENA study web page — http://www.helenastudy.com